CLINICAL TRIAL: NCT00749801
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Comparison Study to Evaluate the Efficacy and Safety of Oral Administration of Nattokinase (From GeneFerm Biotechnology Co., Ltd.) Taken by Dyslipidemia Patients
Brief Title: Efficacy and Safety of Geneferm Nattokinase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi Mei Medical Hospital (Other)
Collaborators: GeneFerm Biotechnology Co., Ltd. (Industry)
Responsible Party: Nae-Cherng Yang, Chungchou Institute of Technology, Changhua, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Geneferm-N01
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Hyperlipidemia
Keywords: drug naive; Dyslipidemic; nattokinase; fibrinolytic
MeSH Terms: conditions — Hyperlipidemias | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): nattokinase-mono formula (3500FU)
  Interventions: Drug: Nattokinase
- B (Experimental): Nattokinase compound-multiple formulae
  Interventions: Drug: Nattokinase
- C (Placebo Comparator): Placebo
  Interventions: Drug: Nattokinase

INTERVENTIONS:
Drug: Nattokinase — 2 capsules in the morning and before bed-time daily
  Other Names: nattokinase-mono formula (3500FU); Nattokinase compound-multiple formulae; Placebo

SUMMARY:
Nattokinase, first found by Dr. Hiroyuki Sumi in 1980, is a potent fibrinolytic enzyme extracted from Natto, a popular soybean fermented food in Japan. It was confirmed that oral administration of nattokinase (or natto) produced a mild and frequent enhancement of the fibrinolytic activity in the plasma as indicated by the fibrinolytic parameters and the production of tissue plasminogen activator. Other studies also showed a reduction in lipid peroxidation and improvement of lipid metabolism. Short-term effect (less then 10 days) of oral administration of nattokinase on both animal and human subjects has been studied and reported. However, whether nattokinase possesses a beneficial effect to dyslipidemic patients remains unclear. The aim of this study is to investigate the long-term effect (six month) of the mono and multiple formulae of nattokinase, change of BP, lipid and fibrinolytic factors from baseline and 6 months on dyslipidemic patients.

DETAILED DESCRIPTION:
This study will employ a randomized, double-blind, placebo-controlled, parallel-group design. Adult men and women who met the inclusion/exclusion criteria and gave consent to participate were randomly assigned to one of the three groups: Group A: nattokinase-mono formula (18 subjects); Group B: nattokinase compound (multiple formulae) (18 subjects); Group C: placebo (10 subjects).

Laboratory tests, including TG, total cholesterol, LDL-C, HDL-C, fibrinogen, D-Dimer, uric acid, vital signs and body weight will be evaluated at screening visit, 1 month, 3 months, 6 months visits after the initiation of treatment. Vital signs and body weight will be measured at every visits.

Patient self-evaluation of tolerance and physical improvement will be assessed by a Patient Questionnaire at each visit. Each patient will be carefully monitored for the development of any adverse events (AE).

The change of all lab tests and vital signs will be plotted and compared against time. Wilcoxon Signed-Rank test will be performed to compare the baseline and 6 months after the initiation of administration. Change from baseline for all lab and vital evaluations will be compared among three groups by Analysis of Variance (ANOVA) followed by LSD multiple comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women above 40 years of age.
2. Dyslipidemic currently being untreated with lipid-lowering drugs. Dyslipidemia is defined as: Total cholesterol 200~300 mg/dl; or Triglyceride 200~500 mg/dl; or Low density lipoprotein-cholesterol 130~200 mg/dl; or High density lipoprotein cholesterol <40 mg/dl (male) and <50 mg/dl (female).
3. Subjects who are, in the opinion of the Investigator, able to comply with the requirements of the study.
4. Subjects who have been adequately informed of the nature and risks of the study and who have given written informed consent prior to receiving investigational product.

Exclusion Criteria:

1. Receipt of lipid-lowering drugs or device within 12 weeks.
2. Myocardial infarction within the preceding 12 weeks.
3. Recent major trauma (within 12 weeks).
4. Recent surgery requiring anesthesia including coronary artery bypass graft (within 12 weeks).
5. Recent hospitalization (within 12 weeks).
6. Acute infection requiring current antibiotic therapy.
7. Recent or abrupt change (within 1 month) in usual diet.
8. Unstable medical condition or life expectancy less than 6 months.
9. Known allergies to the component of study product.
10. Patients have acute disease, and in the opinion of investigators, are not suitable to participate in this study.
11. Total cholesterol >300 mg/dl; or Triglyceride >500 mg/dl; or Low density lipoprotein-cholesterol >200 mg/dl.
12. Current use of warfarin.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Fibrinogen, FDP (fibrin degradation product), D-dimer, Total cholesterol, LDL-C (Low-density lipoprotein cholesterol), HDL-C (High-density lipoprotein cholesterol), Triglyceride (TG), and Uric acid | screening, day 0, weeks 4, 13, 26

SECONDARY OUTCOMES:
Vital signs and self-evaluated questionnaire | screening, day 0, weeks 4, 13, 26

CONTACTS AND LOCATIONS:
Overall Officials: Nae-Cherng Yang, PhD, Study Chair — Chung Chou Institute of Technology
Locations (1):
- Chi Mei Medical Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Yang NC, Chou CW, Chen CY, Hwang KL, Yang YC. Combined nattokinase with red yeast rice but not nattokinase alone has potent effects on blood lipids in human subjects with hyperlipidemia. Asia Pac J Clin Nutr. 2009;18(3):310-7. PMID 19786378